CLINICAL TRIAL: NCT02781337
Title: Epidemiological and Molecular Colorectal Cancer Registry
Acronym: EMR-CRC
Status: Recruiting | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Carlos Vaccaro, MD, Hospital Italiano de Buenos Aires
Other Study IDs: 1513; REM-CCR (Registry Identifier: Epidemiological and Molecular Colorectal Cancer Registry)
Record Dates: First submitted 2016-05-17; First posted 2016-05-24 (Estimated); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Neoplasms; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Tissue samples and blood specimens are frozen and store at Eighty degrees below 0 degrees Celsius (-80ºC).
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a Registry that invites patients undergoing colorectal surgery for colorectal cancer. Epidemiological data is collected. The Registry includes tumor tissue and blood banks for analyzing different genetic mutations and disease-specific biomarkers.

DETAILED DESCRIPTION:
This is a Registry that invites patients undergoing colorectal surgery for colorectal cancer. Epidemiological data is collected. The Registry includes tumor tissue and blood samples banks used to studied different genetic variants and disease-specific biomarkers present in patients with Lynch syndrome and others hereditary cancers.

The aim of this registry is to set up the necessary resources to help basic and clinical research projects on colorectal cancer (CRC) within the Hospital Italiano de Buenos Aires (HIBA) and promote scientific collaborations between the HIBA and other institutions within and outside the country.

To make this project, the following specific goals are proposed:

Objective 1: Establishment of an efficient algorithm to enroll patients diagnosed with CRC from HIBA, through collaboration between the services of Surgery, Gastroenterology, Pathology, Oncology, Institute of Translational Medicine and Biomedical Engineering (IMTIB), Medical Clinic and Medical Informatics.

Objective 2: Development of logistics for the connection and expansion of the bank of biological samples (DNA, serum) and tumor samples (tissue fixed in formalin, frozen tissue) to the CRC.

Objective 3: Development of computer software to record data about patient enrolled in a dynamic way.

Objective 4: Development of pipelines and create a supervisory committee to regulate the future of samples and data obtained through the registry, accord the current standards of ethical code, and improve the current collaborations with foreign researchers.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing colorectal surgery for colorectal cancer.

Exclusion Criteria:

* Unwillingness to participate.

Ages: 21 Years to 96 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing colorectal surgery due to colorectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 2100 (Estimated)
Dates: Start 2012-05; Primary Completion 2027-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Patient overall survival at 5 years.
Disease-free survival | 5 years
  The time free of disease recurrence will be estimated in the whole cohort and according to colorectal cancer stages and molecular profiles.

SECONDARY OUTCOMES:
Molecular characteristics of colorectal adenocarcinoma. | 0
  At initial diagnosis, molecular tumor markers will be determined in the tissue samples.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Vaccaro, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, CABA, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Collura A, Lagrange A, Svrcek M, Marisa L, Buhard O, Guilloux A, Wanherdrick K, Dorard C, Taieb A, Saget A, Loh M, Soong R, Zeps N, Platell C, Mews A, Iacopetta B, De Thonel A, Seigneuric R, Marcion G, Chapusot C, Lepage C, Bouvier AM, Gaub MP, Milano G, Selves J, Senet P, Delarue P, Arzouk H, Lacoste C, Coquelle A, Bengrine-Lefevre L, Tournigand C, Lefevre JH, Parc Y, Biard DS, Flejou JF, Garrido C, Duval A. Patients with colorectal tumors with microsatellite instability and large deletions in HSP110 T17 have improved response to 5-fluorouracil-based chemotherapy. Gastroenterology. 2014 Feb;146(2):401-11.e1. doi: 10.1053/j.gastro.2013.10.054. PMID 24512910
- [Background] Kim JH, Kang GH. Molecular and prognostic heterogeneity of microsatellite-unstable colorectal cancer. World J Gastroenterol. 2014 Apr 21;20(15):4230-43. doi: 10.3748/wjg.v20.i15.4230. PMID 24764661
- [Background] Phipps AI, Limburg PJ, Baron JA, Burnett-Hartman AN, Weisenberger DJ, Laird PW, Sinicrope FA, Rosty C, Buchanan DD, Potter JD, Newcomb PA. Association between molecular subtypes of colorectal cancer and patient survival. Gastroenterology. 2015 Jan;148(1):77-87.e2. doi: 10.1053/j.gastro.2014.09.038. Epub 2014 Sep 30. PMID 25280443
- [Background] Kim JH, Bae JM, Oh HJ, Lee HS, Kang GH. Pathologic Factors Associated with Prognosis after Adjuvant Chemotherapy in Stage II/III Microsatellite-Unstable Colorectal Cancers. J Pathol Transl Med. 2015 Mar;49(2):118-28. doi: 10.4132/jptm.2015.02.05. Epub 2015 Mar 12. PMID 26148739
- [Background] Jenkins MA, Hayashi S, O'Shea AM, Burgart LJ, Smyrk TC, Shimizu D, Waring PM, Ruszkiewicz AR, Pollett AF, Redston M, Barker MA, Baron JA, Casey GR, Dowty JG, Giles GG, Limburg P, Newcomb P, Young JP, Walsh MD, Thibodeau SN, Lindor NM, Lemarchand L, Gallinger S, Haile RW, Potter JD, Hopper JL, Jass JR; Colon Cancer Family Registry. Pathology features in Bethesda guidelines predict colorectal cancer microsatellite instability: a population-based study. Gastroenterology. 2007 Jul;133(1):48-56. doi: 10.1053/j.gastro.2007.04.044. Epub 2007 Apr 25. PMID 17631130
- [Background] Webber EM, Kauffman TL, O'Connor E, Goddard KA. Systematic review of the predictive effect of MSI status in colorectal cancer patients undergoing 5FU-based chemotherapy. BMC Cancer. 2015 Mar 21;15:156. doi: 10.1186/s12885-015-1093-4. PMID 25884995
- [Background] Park JG, Kim DW, Hong CW, Nam BH, Shin YK, Hong SH, Kim IJ, Lim SB, Aronson M, Bisgaard ML, Brown GJ, Burn J, Chow E, Conrad P, Douglas F, Dunlop M, Ford J, Greenblatt MS, Heikki J, Heinimann K, Lynch EL, Macrae F, McKinnon WC, Moeslein G, Rossi BM, Rozen P, Schofield L, Vaccaro C, Vasen H, Velthuizen M, Viel A, Wijnen J; International Society for Gastrointestinal Hereditary Tumours. Germ line mutations of mismatch repair genes in hereditary nonpolyposis colorectal cancer patients with small bowel cancer: International Society for Gastrointestinal Hereditary Tumours Collaborative Study. Clin Cancer Res. 2006 Jun 1;12(11 Pt 1):3389-93. doi: 10.1158/1078-0432.CCR-05-2452. PMID 16740762
- [Background] Jass JR. Classification of colorectal cancer based on correlation of clinical, morphological and molecular features. Histopathology. 2007 Jan;50(1):113-30. doi: 10.1111/j.1365-2559.2006.02549.x. PMID 17204026